CLINICAL TRIAL: NCT00737503
Title: Introduction of an Oral Live Human Rotavirus (Rotarix) Vaccine in Matlab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: PATH (Other)
Responsible Party: DR. K. ZAMAN, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-024
Record Dates: First submitted 2008-08-16; First posted 2008-08-19 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2008-08

CONDITIONS: Rotavirus Gastroenteritis
Keywords: vaccine effectiveness, rotavirus, diarrhoea, Bangladesh
MeSH Terms: conditions — Diarrhea | interventions — Rotavirus Vaccines; RIX4414 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): All eligible children in the experimental arm will be vaccinated with the Rotavirus vaccine
  Interventions: Biological: Rotavirus Vaccine (ROTARIX)
- 2 (No Intervention): Children will not be vaccinated with rotavirus vaccine.

INTERVENTIONS:
Biological: Rotavirus Vaccine (ROTARIX) — Rotavirus Vaccine two doses four weeks apart
  Other Names: ROTARIX
  Arms: 1

SUMMARY:
The study will be conducted in the Matlab Health and Demographic Surveillance System (HDSS) field area of the International Centre for Diarrhoeal Disease Research, Bangladesh (ICDDR,B) to determine the population effectiveness of Rotarix in Bangladeshi children. Villages in both intervention and government comparison areas will be included in this evaluation. We propose to introduce Rotarix into half of the villages of the Matlab HDSS. In villages randomized to receive the vaccine, all eligible children will be offered Rotarix during their first two Expanded Programme on Immunization (EPI) visits, as would routinely be done if Rotarix were included in the Government EPI schedule. In villages randomized not to receive Rotarix, children will receive their EPI vaccinations exactly as they would have in the absence of this study. Administration of Rotarix will be conducted by regular EPI staff, but ICDDR,B study staff will be present to document informed consent and collect study-specific information. The Ministry of Health will be an active partner in this evaluation since they will be the agency which may follow up with any subsequent vaccine programme. Vaccination with Rotarix will be recorded on the infant's immunization card which is normally used by the EPI programme, but also on a separate study-specific data collection form.

Vaccination with Rotarix will continue from study initiation through June 30, 2011. Surveillance for rotavirus gastroenteritis will occur at Matlab Diarrhoeal Hospital and the community treatment centres of the Matlab HDSS continuously throughout the study period. Diarrheal illness information collected through surveillance will be linked to Rotarix study-specific data through the subject's HDSS identification numbers. The primary study endpoint will be the occurrence of an illness episode of acute diarrhoea, among infants and children admitted to a medical facility, determined to be caused by wild-type rotavirus found in a stool specimen. At the end of the surveillance period, rates of this primary study endpoint among age-eligible infants will be compared for villages randomized to receive Rotarix versus for villages randomized not to receive Rotarix. We expect that the rates of rotavirus diarrhoea will be significantly lower among children from the vaccinated villages.

The first participant was enrolled in the study on September 23, 2008. Till date (May 12, 2010) a total of 2,882 participants have been enrolled and received first dose. 2,684 participants received second dose of Rotarix. There were 1013 cases gastroentritis reported to diarrhoeal treatment centres among <2 years old children from the vaccinated and unvaccinated villages. There were six death cases among the children who received Rotarix vaccine. These death cases were not related to the vaccines/study products.

DETAILED DESCRIPTION:
This trial will determine the population effectiveness of Rotarix in Bangladeshi infants. The study will be conducted in both the government comparison area and the intervention area of the Matlab HDSS. To carry out the evaluation, we will introduce the Rotarix vaccine into half of the villages of the HDSS area. In villages randomized to receive Rotarix, the study will be explained to parents and if they consent to their child's participation and the child is eligible, the child will receive two doses of Rotarix during their first two EPI visits (scheduled for 6 and 10 weeks of age), if possible, as would routinely be done if Rotarix were included in the government programme. Administration of Rotarix will be conducted by regular EPI staff, but ICDDR,B study staff will be present to document informed consent and collect study-specific information. Vaccination with Rotarix will be recorded on the infant's immunization card which is normally used by the EPI programme, but also on a separate study-specific data collection form. Participation in the study will not affect a subject's receipt of other routine childhood immunizations or other medical care. In villages randomized not to receive Rotarix, children will receive their EPI vaccinations exactly as they would have in the absence of this study.

Surveillance for will be conducted at the Matlab Diarrhoeal Hospital and the two community treatment centres at Nayergaon and Kalirbazaar, which facilitate quick and easy accessibility of treatment for life-threatening diarrhoeal diseases from the HDSS area. The main study outcome will be episodes of rotavirus diarrhoea among children admitted to Matlab Diarrhoeal Hospital or either of the two community treatment centres (Nayergaon and Kalirbazaar). Study personnel will record the child's symptoms and clinical history, and collect a fecal specimen for laboratory testing for rotavirus. The identity of the child will be confirmed through the HDSS subject identification number system. All patients coming to the Matlab Diarrhoea Hospital and Nayergoan community treatment centre from these villages are already included in the Matlab diarrhoea surveillance system, and faecal samples are routinely tested for rotavirus and other pathogens, with results linked to demographic and health databases of the HDSS. Kalirbazaar treatment centre is not currently included in the current surveillance system, but we will establish surveillance at this centre during this study. For enrolled participants who present to one of the treatment facilities, illness information and test results will be linked to HDSS demographic data and study-specific data collected at enrolment through the subject's HDSS number. For residents not enrolled who present to a treatment facility, illness information will be linked only to HDSS demographic data, as is already being done as part of surveillance activities.

Rates of acute gastroenteritis caused by rotavirus and other agents among age-eligible infants will be compared for infants (vaccinated and unvaccinated) from villages randomized to receive Rotarix versus for those (unvaccinated) from villages randomized not to receive Rotarix. We expect that the rates of diarrhoea will be significantly lower among children from the vaccinated villages, but that rates of diarrhoea caused by other pathogens may be similar. (This second analysis - a "control analysis" - will be helpful to verify a lack of bias in health seeking behaviours since one would expect that cholera, ETEC, Salmonella and Shigella gastroenteritis rates would be similar in the two groups.). These cases will be detected from all patients of all ages who come to the Matlab Diarrhoeal Hospital or the community treatment centres (Nayergaon or Kalirbazaar), but the primary analysis will include only those rotavirus diarrhoea cases among children who had been age-eligible for vaccination in their respective villages.

Although not a blinded evaluation, the introduction of bias will be reduced in several ways. First, the vaccine teams located in the EPI centres that are completely separate from the clinical settings where clinicians will be conducting surveillance. Second, the clinicians are separated from those scientists conducting laboratory testing. Third, laboratory assays for rotavirus will be carried out in the laboratory in Dhaka using coded specimens and are not conducted at the time of illness (since they have little clinical value). Although a parent could inform the clinician as to his/her child's participation in the study, this is believed to be an unlikely or important source of bias for two reasons. One, most rotavirus gastroenteritis is not seen until later than 6 months after an infant's second dose of Rotarix, and there will be no active follow-up among parents after last receipt of Rotarix. Thus, there is a reduced likelihood that parents will remember that their child had received a vaccination targeted specifically against one type of severe diarrhoea. Second, Matlab Diarrhoeal Hospital and the community treatment centres have been caring for severe diarrhoea for many years and the entire community is already accustomed to attending the facilities for such illnesses. Thus, there is a reduced likelihood parents of vaccinated and unvaccinated infants are going to have differential diarrhoeal illness treatment-seeking behaviors.

Again, the study will be conducted in both the government comparison area and the intervention area of Matlab HDSS. Enrolment will begin in the government comparison area no later than June 1, 2008. Enrolment will begin in the intervention area January 1, 2009. Surveillance for rotavirus diarrhoea will occur continuously and concurrently to enrolment activities. Enrolment in both areas will cease on June 30, 2010, but surveillance for rotavirus gastroenteritis will occur until December 31, 2010.

By in January 1, 2009, it is expected that less than 15% of children less than 2 years of age in the intervention area will have received Rotateq in the Merck trial. Nonetheless, we will stratify randomization within the intervention area by rates of participation in that trial for each village. Additionally, because we will have the full dataset for Matlab for the Rotateq trial, we will be able to analyze any impact of that Rotateq trial on the Rotarix evaluation within the intervention area.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant at least 6 weeks of age and not older than 20 weeks of age at the time of first dose of Rotarix.
* An infant whose parent or guardian's primary residence, at the time of first EPI vaccinations, is a village selected to receive Rotarix.
* Written informed consent obtained from the parent or guardian of the subject, prior to the subject's first study vaccination

Exclusion Criteria:

* Hypersensitivity to the active substance or any component in the vaccine
* Hypersensitivity after previous administration of rotavirus vaccines.
* Previous history of intussusception.
* Subjects with uncorrected congenital malformation of the gastrointestinal tract that would predispose for intussusception.
* Infants with known or suspected immunodeficiency.
* Administration of Rotarix should be postponed in subjects suffering from an acute severe febrile illness only if that illness also results in postponement of other EPI vaccinations.

Ages: 6 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4550 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Primary study endpoint: acute rotavirus diarrhoea occurring from 6 weeks of age to the end of the follow-up period in subjects who resided in randomized villages during the period when they were age-eligible to have received Rotarix. | 24 months

SECONDARY OUTCOMES:
Rates of all cause acute diarrhoea | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Zaman K, Sack DA, Neuzil KM, Yunus M, Moulton LH, Sugimoto JD, Fleming JA, Hossain I, Arifeen SE, Azim T, Rahman M, Lewis KDC, Feller AJ, Qadri F, Halloran ME, Cravioto A, Victor JC. Effectiveness of a live oral human rotavirus vaccine after programmatic introduction in Bangladesh: A cluster-randomized trial. PLoS Med. 2017 Apr 18;14(4):e1002282. doi: 10.1371/journal.pmed.1002282. eCollection 2017 Apr. PMID 28419095